CLINICAL TRIAL: NCT01641107
Title: Front-line Treatment of Philadelphia Positive/BCR-ABL Positive Acute Lymphoblastic Leukemia With Ponatinib, a New Potent Tyrosine Kinase Inhibitor.
Brief Title: Phase II Front-line Ponatinib in Adult Philadelphia+/BCR-ABL+ Acute Lymphoblastic Leukemia.
Acronym: LAL1811
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1811; 2012-002761-35 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Philadelphia Positive; BCR-ABL Positive; Acute Lymphoblastic Leukemia
Keywords: Ph+; BCR-ABL+; ALL; Ponatinib; stem cell transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ponatinib (Experimental)
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Treatment:
  Patients will receive daily oral administration of Ponatinib at a dose of 45 mg/day for 6 weeks (defined as one course) for 8 courses, same dose and schedule, for a total of 48 weeks. Each patient will be followed for the subsequent 24 months, every 3 month, providing survival information and monitoring serious adverse event. Each patient should be treated for a minimum of 6 weeks. Patients must be discontinued from the trial in the event of myocardial infarction or stroke, or for development or progression of arterial disease necessitating revascularization. Once a complete hematologic response has been achieved, with a platelet count ≥ 50x109/L, patients can be treated with aspirin and/or a statin as clinically indicated, at investigator discretion.

SUMMARY:
Drug resistance resulting from emergence of Imatinib-resistant BCR-ABL clones is a significant problem in Ph positive ALL patients because after a very good initial response to one TKI inhibitor, many patients relapse within one year, relapse being almost always associated with a BCR-ABL kinase domain point mutation. The patients who relapse after treatment with one TKI can be rescued to remission with another TKI, but the second remission is usually shorter than the previous one. A more potent TKI inhibitor, and pan-active not only on all the BCR-ABL variants (including the second generation TKI resistant T315I mutant), but also on others molecular targets can do better. In this context, Ponatinib is a novel synthetic orally active tyrosine kinase inhibitor (TKI), specifically developed to inhibit BCR-ABL, the fusion protein that is the product of the Philadelphia chromosome (Ph) in chronic myeloid leukemia (CML) and in a subset of acute lymphoblastic leukemia (Ph+ ALL). It potently inhibits the BCR-ABL protein as well as mutated forms of the protein that arise in patients resistant to prior therapies with TKIs. Ponatinib has been demonstrated to inhibit all the mutations that have been detected so far, in vitro and in vivo and to uniformly suppress the emerge of single-mutant clones in a mutagenesis assay. In the Phase II study, 41% of Philadelphia chromosome positive acute lymphoblastic leukemia patients treated with Ponatinib achieved major hematologic response, 47% had a major cytogenetic response, 38% obtained a complete cytogenetic response, showing that Ponatinib provides significant benefit despite previous intolerance or refractoriness to other TKIs. The Phase I trial showed that patients with a more recent diagnosis had increased rates of major molecular response: 79% for 14 patients with 0 to 5 years since diagnosis vs. 29% for 14 patients with more than 5 to 9 years since diagnosis (P=0.02) and 27% for 15 patients with more than 9 to 24 years since diagnosis (P=0.009). These characteristics support the hypothesis for a role of Ponatinib not only in patients resistant to prior TKI therapy but also in untreated ALL Ph+ patients, in order to prevent the emergence of resistant caused by the selection of mutated Ph+ clones and in order to avoid rapid progression of the disease.

DETAILED DESCRIPTION:
This is a multi-center, phase 2, single arm unblinded trial of oral Ponatinib in patients with Ph+ Acute Lymphoblastic Leukemia. Patients will receive daily oral administration of Ponatinib at a dose of 45 mg/day for 6 weeks (defined as one course) for 8 courses, same dose and schedule, for a total of 48 weeks. Each patient will be followed for the subsequent 24 months, every 3 month, providing survival information and monitoring serious adverse event.

Each patient should be treated for a minimum of 6 weeks. Then a patient can be discontinued in the following situation:

* at the end of first course (6 weeks), in case of lack of CHR;
* at the end of third course (18 weeks), in case of lack of CCgR;
* any time in case of loss of CHR or CCgR.

If they remain on therapy after 48 weeks, they will be able to continue treatment during the extension phase of the study, if it is of interest of the patient, or they will be allowed to receive any treatment that is in their interest. For all the patients remaining on trial, response, outcome and toxicity will be followed for the subsequent 24 months.The 6-weeks periodicity must be rigidly respected, irrespective of the temporary discontinuation of study drug (eg, if a patient will take Ponatinib only for 4 weeks and will remain off-treatment for the subsequent two weeks because of AE, when the 7th week begins this patient will restart Ponatinib as a second course, as per protocol). Prednisone (P) will be administered to all patients for 7-14 days, before Ponatinib, so as to make it possible to wait for the results of cytogenetic and molecular tests, and to evaluate the response to P alone, hence for another 21 days. Intrathecal therapy (IT) with MTX/AraC/DEX is mandatory, every 28 days, in patients without clinical-cytologic evidence of meningeal involvement. In patients with CNS disease, IT is performed twice weekly until a complete clearance of cerebrospinal fluid blast cells is achieved, hence once weekly for 4 weeks, hence once monthly.

ELIGIBILITY:
Inclusion Criteria:

1. To be classified as having Ph+ ALL, patients must have >20% blasts in bone marrow at the time of diagnosis and no prior history of CML.
2. Patients with previously untreated Ph+ and/or BCR/ABL + ALL:

   * age ≥ 60 years old or
   * age ≥ 18 years old, but unfit for program of intensive therapy and allogeneic SCT
3. Adequate hepatic function as defined by the following criteria:

   * total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome
   * alanine aminotransferase (ALT) ≤2.5 × ULN
   * aspartate aminotransferase (AST) ≤2.5 × ULN.
4. Adequate pancreatic function as defined by the following criterion:

   - serum lipase and amylase ≤1.5 × ULN.
5. For females of childbearing potential, a negative pregnancy test must be documented prior to randomization.
6. Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from randomization through 4 months after the end of treatment.
7. Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

1. WHO performance status ≤ 50% (Karnofsky) or ≥ 3 (ECOG).
2. Active HBV or HCV hepatitis, or AST/ALT ≥ 2.5 x ULN and bilirubin ≥ 1.5 x ULN.
3. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis.
4. History of alcohol abuse.
5. Ongoing or active infections.
6. Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
7. Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   * any history of myocardial infarction, stroke, or revascularization
   * unstable angina or transient ischemic attack within 6 months prior to enrollment
   * congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards within 6 months prior to enrollment
   * history of clinically significant (as determined by the treating physician) atrial arrhythmia
   * any history of ventricular arrhythmia
   * any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism .
8. Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
9. Taking medications that are known to be associated with Torsades de Pointes.
10. Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
11. Creatinine level > 2.5mg/dl or Glomerular Filtration Rate (GFR) < 20 ml/min or proteinuria > 3.5 g/day.
12. Impairment of gastrointestinal (GI) function, or a GI disease that may significantly alter the absorption of study drugs (e.g. rare hereditary problems of galactose intolerance , the Lapp lactase deficiency or glucose-galactose malabsorption, severe malabsorption syndrome, or extended small bowel resection).
13. Patients who are currently receiving treatment with any of the medications listed in Appendix E if the medications cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in Appendix E have the potential to prolong QT.
14. Patients who have received any investigational drug ≤ 4 weeks.
15. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
16. Patients who are pregnant or breast feeding and adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of Ponatinib). Post menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 4 months following discontinuation of study drugs.
17. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
18. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are in Complete Hematological Response (CHR). | At 6 months from study entry.
  The primary endpoint is the proportion of patients who are in CHR at 6 months, calculated on the total number of patients who have been enroled and have received at least one dose of the first drug (prednisone).

SECONDARY OUTCOMES:
The rate of Complete Hematological Response (CHR). | At 6, 12, 24, 36 and 48 weeks from study entry.
  CHR requires that all of the following are present:
  * Bone marrow with less than 5% blast cells
  * Peripheral blood differential without blasts
  * PMN ≥ 1.5 x 109/L
  * PLT ≥ 100 x 109/L
  * No evidence of extramedullary involvement from leukemia
The rate of complete Cytogenetic Response (CgR). | At 6, 12, 24, 36 and 48 weeks from study entry.
  CgR is defined based on the percentage of Ph pos metaphases, as evaluated by chromosome banding analysis (CBA) of at least 20 marrow cell metaphases:
  1. Complete (CCgR) if Ph pos 0
  2. Partial (PCgR) if Ph pos 1-34%
  3. Minor (mCgR) if Ph pos 35-65%
  4. Minimal or none (min/none CgR) if Ph pos > 65% If only interphase FISH data are available, the response can be defined only as non-complete or complete - to be complete by FISH, it is required that less than 1% of nuclei (minimum number 200) have a positive signal.
Duration of Complete Cytogenetic Response (CCgR). | After four years from study entry.
  Duration of CCgR is measured by the date of the achievement of CCgR to the date of CCgR loss.
The rate of Complete Molecular Response (CMoIR). | At 12, 24, 36 and 48 weeks from study entry.
  Molecular response is classified as:
  • Complete if by RT-Q-PCR the BCR-ABL: ABL ratio is below 0.01, with a sensitivity of at least 30,000 molecules of ABL.
The rate of major molecular response. | At 12, 24, 36 and 48 weeks from study entry.
  Molecular response (MR) is classified as:
  • Major (MMolR) if by RT-Q-PCR the BCR-ABL: ABL ratio is lower than 0.10, with a sensitivity of at least 30,000 molecules of ABL.
Duration of Complete molecular response (CMR). | After four years from study entry.
  Duration of CMR is measured by the date of the achievement of CMR to the date of CMR loss.
Type and number of BCR-ABL kinase domain mutations. | At the end of the study. At four years after enrollment of first patient.
Percentage of relationships between the response and the biomarkers. | At six months from study entry.
Event Free Survival. | After four years from study entry.
  Events are induction failure, relapse and death whichever comes first.
Overall survival | At the end of study. After four years from enrolment.
  Overall survival is measured in all patients from the data of enrolment to the date of death, by any causes.
Failure Free Survival | After four years from study entry.
Rate of Rate of side effects, adverse events and serious adverse events. | After four years from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, Pr., Principal Investigator — Dpt of Hematology and Oncology "Seràgnoli", "Sant'Orsola-Malpighi" University Hospital of Bologna
Locations (42):
- Italy (42):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - Dipartimento Area Medica - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Ferrara
  - Policlinico di Careggi, Florence
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Unità Operativa Complessa - Medicina Generale - Sezione di Ematologia - Ospedale Versilia USL 12 Toscana, Lido di Camaiore
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - Ospedale Niguarda " Ca Granda", Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvator, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Ospedale "Infermi", Rimini
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - UOC di Ematologia e Trapianti di Cellule Staminali Emopoietiche - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Azienda U.L.S.S.9 - U.O. di Ematologia, Treviso
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza

REFERENCES:
- [Derived] Martinelli G, Papayannidis C, Piciocchi A, Robustelli V, Soverini S, Terragna C, Marconi G, Lemoli RM, Guolo F, Fornaro A, Lunghi M, de Fabritiis P, Candoni A, Selleri C, Simonetti F, Bocchia M, Vitale A, Frison L, Tedeschi A, Cuneo A, Bonifacio M, Martelli MP, D'Ardia S, Trappolini S, Tosi P, Galieni P, Fabbiano F, Abbenante MC, Granier M, Zhu Z, Wang M, Sartor C, Paolini S, Cavo M, Foa R, Fazi P, Vignetti M, Baccarani M. INCB84344-201: Ponatinib and steroids in frontline therapy for unfit patients with Ph+ acute lymphoblastic leukemia. Blood Adv. 2022 Mar 22;6(6):1742-1753. doi: 10.1182/bloodadvances.2021004821. PMID 34649276
- See also: Gimema Foundation Website — http://www.gimema.it